CLINICAL TRIAL: NCT04808544
Title: Efficacy of Preoperative Injection of Naldebain® in Management of Acute and Chronic Pain After Laparoscopic Cholecystectomy
Brief Title: Naldebain for Pain Management of Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMRP28110N
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative; Pain, Chronic; Cholecystitis; Quality of Life
Keywords: Nalbupine; Dinalbuphine sebacate; Naldebain; Opioid; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Cholecystitis | interventions — sebacoyl dinalbuphine ester; benzyl benzoate; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Naldebain (active drug in solvent containing benzyl benzoate and sesame oil) or placebo drug (solvent containing benzyl benzoate and sesame oil) will be prepared by the clinical pharmacists in an identical injection syringe within 30 min before injection. The participants, anesthesiologists, surgeons, investigators and outcomes assessors will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): Patients assigned to placebo group will receive a single intramuscular injection of 2 ml solvent containing benzyl benzoate and sesame oil into the gluteus muscles under ultrasound-guidance.
  Interventions: Drug: Placebo solution
- Naldebain group (Active Comparator): Patients assigned to Naldebain group will receive a single intramuscular injection of dinalbuphine sebacate (150 mg in 2 ml solvent containing benzyl benzoate and sesame oil) into the gluteus muscles under ultrasound-guidance.
  Interventions: Drug: Dinalbuphine sebacate

INTERVENTIONS:
Drug: Dinalbuphine sebacate — Naldebain dissolved in benzyl benzoate and sesame oil (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance.
  Other Names: Naldebain ER®; Sebacoyl Dinalbuphine Ester Injection
  Arms: Naldebain group
Drug: Placebo solution — Benzyl benzoate and sesame oil served as placebo solution (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance.
  Other Names: Benzyl benzoate and sesame oil
  Arms: Placebo group

SUMMARY:
Laparoscopic cholecystectomy is the most common surgical procedure for removal of the inflamed gall bladder or other gall bladder pathologies. There are more than 12,000 cases of cholecystectomy performed in Taiwan annually, and more than 85% of this procedure are undertook with laparoscopic techniques. Even with minimally invasive laparoscopic operation, patients may still suffer from postoperative wound pain, deep visceral or referred pain. About 80% of patients who received laparoscopic procedures complain of moderate-to-severe pain within the first day after cholecystectomy. Most importantly, up to 20% (range from 3 to 20%) of these patients complained surgical-related pain one year after operation and they require prolonged use of opioid to control chronic postoperative pain (CPSP). However, there are currently lack of clinical practice guidelines or recommendations for prevention of CPSP after laparoscopic abdominal surgery. Although regional block techniques (i.e. truncal block or intrathecal opioid) are considered as effective supplementary analgesic approaches to improve postoperative pain control, parenteral administration of analgesics remain as the mainstay for pain management of laparoscopic abdominal surgery. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is an extended-release dinalbuphine sebacate, and is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. A number of clinical studies have shown that single-dose of pre-operative intramuscular administration of Naldebain® provides significantly higher analgesic effect up to 1 week in hemorrhoidectomy and laparotomy surgery with a well-tolerated safety profile. Therefore, this PI-initiated randomized, double-blind, placebo-control trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in patients receiving laparoscopic cholecystectomy, and prevention of the development of CPSP after surgery.

DETAILED DESCRIPTION:
Clinical studies indicate that more than 80% of patients suffer from surgical-related pain in the first few days after major laparotomy or laparoscopic abdominal surgery and about 10% of these patients may develop chronic postoperative pain (CPSP), which can last up to several years after surgery. One of the major risk factors for developing CPSP is inadequate management of the acute postoperative pain. Laparoscopic cholecystectomy is the most common surgical procedure for removal of the inflamed gall bladder or other gall bladder pathologies. There are more than 12,000 cases of cholecystectomy performed in Taiwan annually, and more than 85% of this procedure are undertook with laparoscopic techniques. Even with the minimally invasive laparoscopic operation, patients may still suffer from acute postoperative surgical-related pain. About 80% of patients who received laparoscopic procedures complain of moderate-to-severe pain within the first day after cholecystectomy. Most importantly, up to 20% (range from 3 to 20%) of these patients complained surgical-related pain one year after operation and they require prolonged use of opioid to control CPSP. The proposed mechanisms of CPSP after laparoscopic cholecystectomy include somatic component (incisional wound pain), visceral component (deep abdominal pain) and referred pain component (shoulder pain). Several important clinical observational studies suggested that inadequate management of surgical-related pain within one week after cholecystectomy is one of the major risk factors for developing CPSP. In addition to pain-related complications, CPSP may also impair patient's quality of life after surgery. However, there are currently lack of clinical practice guidelines or recommendations for prevention of CPSP after laparoscopic abdominal surgery. Although regional block techniques (i.e. truncal block or intrathecal opioid) are considered as effective supplementary analgesic approaches to improve postoperative pain control, parenteral administration of analgesics remain as the mainstay for pain management of laparoscopic abdominal surgery. Nalbuphine is a semi-synthetic opioid that acts as a mixed kappa opioid agonist and mu opioid antagonist, but its clinical applications in relieving acute postoperative pain is limited by the relatively short duration of action of 3-6h. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is an extended-release dinalbuphine sebacate, and is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. A number of clinical studies have shown that single-dose of pre-operative intramuscular administration of Naldebain® provides significantly higher analgesic effect up to 1 week in hemorrhoidectomy and laparotomy surgery with a well-tolerated safety profile. Naldebain® has not been tested in laparoscopic surgery. Therefore, this PI-initiated randomized, double-blind, placebo-control trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in patients receiving laparoscopic cholecystectomy, and prevention of the development of CPSP after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to receive laparoscopic cholecystectomy

Exclusion Criteria:

* Emergency operation
* Open cholecystectomy
* American Society of Anesthesiologists physical status > or =4
* Chronic opioid user
* Allergy to nalbuphine, benzyl benzoate or sesame oil
* Anticipated to receive ventilator support via an endotracheal tube after operation
* Unable for verbal pain assessment or not able to participate questionnaire survey

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain | 7 days after surgery
  Pain score measured by visual analogue scale (VAS 1-10, a continuum scale in which 0 represents "no pain" and and 10 represents "worst pain.")
Total requirement dose of rescue analgesics | 7 days after surgery
  Total doses of opioids, NSAIDs, COX-2 inhibitors administered

SECONDARY OUTCOMES:
Incidence of chronic post-surgical pain | 3 months after surgery
  Pain that newly develops after operation and lasts >2 months and other causes of pain are excluded
Quality of life after surgery | 3 months after surgery
  Quality of life will be assessed by the HRQoL SF -12 Questionnaire, which consists a physical component summary (PCS) and a mental component summary (MCS). The rating scales range from yes-no to likert scales, and the final score of PCS and MCS will be calculated by an algorithm (QualityMetric's SF-12v1®). Scores range from 0 to 100, in which lower scores mean lower health related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da Hospital, Yanchao, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No